CLINICAL TRIAL: NCT05674942
Title: Urinary Tract Infection in Patients With Chronic Kidney Disease: A Retrospective Observational Study at Outpatient Nephrology Clinics
Brief Title: Urinary Tract Infection in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Assistant professor & lecturer, Alexandria University
Other Study IDs: Urinary Tract Infection
Record Dates: First submitted 2022-12-14; First posted 2023-01-09 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Urinary Tract Infections; Chronic Kidney Diseases
Keywords: urinary tract; infection; chronic kidney disease; UTI; CKD
MeSH Terms: conditions — Urinary Tract Infections; Renal Insufficiency, Chronic; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with urinary tract infection and chronic kidney disease — The data that will be collected from the electronic patient records at the clinics through a google form will include sociodemographic (age, sex, weight and occupation), comorbidities (e.g., HTN, DM), medications used, renal functions (serum creatinine, and CKD stage calculated by 2021 CKD-EPI creatinine equation), and in case of positive urine culture (type of microorganism and antibiogram).

SUMMARY:
This study aims to investigate the etiology and associated risk factors for UTI in Egyptian chronic kidney disease patients. In addition, to identify the isolated micro-organisms and their sensitivity patterns for better anticipation of treatment regimen.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) patients are at higher risk of urinary tract infections (UTI), as CKD is a state of chronic inflammation, metabolic disturbance and impaired immunocompetence. Moreover, patient with CKD are usually of advanced age and suffer from other comorbidities such as diabetes, hypertension, obesity, and cardiovascular diseases, which also add to their risk of infection.

UTI comprises heterogeneous conditions ranging from mild cystitis, easily treated with oral antibiotics, to life-threatening sepsis and multiple organ failure.

There is scarce information about risk factors of recurrence of UTI and infection with multidrug-resistant organisms in the Egyptian population.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females aged ≥ 18 years old
2. Patients with CKD stages (G1 to G4)
3. Patients diagnosed with UTI due to urine culture

Exclusion Criteria:

1. Non-CKD patients
2. pregnant females
3. CKD patients on immunosuppressant agents
4. ESRD patients on hemodialysis
5. Patients with structural abnormalities which make them liable to frequent UTI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from outpatient nephrology clinics in Alexandria.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
prevalence of UTI in CKD patients | records will be retrospectively screened from January 2019 till September 2022
  percentage of UTI in CKD patients
isolated microorganisms causing UTI in CKD patients | records will be retrospectively screened from January 2019 till September 2022
  isolated microorganisms in cultures causing UTI in CKD patients

SECONDARY OUTCOMES:
sensitivity pattern of urine cultures in CKD | records will be retrospectively screened from January 2019 till September 2022
  describe sensitivity pattern of urine cultures in CKD

CONTACTS AND LOCATIONS:
Overall Officials: mohamed mamdouh elsayed, MD, Principal Investigator — Lecturer of Nephrology & Internal Medicine, Faculty of medicine, Alexandria University; Mohammed Abdel Gawad, Study Chair — Nephrology Lecturer, School of Medicine, New Giza University (NGU), Giza, Egypt; Dalia Elzayat, Study Chair — Faculty of Pharmacy, Pharos University, Alexandria, Egypt; Reham Mekawy, Study Chair — Faculty of Pharmacy, Pharos University, Alexandria, Egypt; Salma Mahdy, Study Chair — Faculty of Pharmacy, Pharos University, Alexandria, Egypt; Salma Imam, Study Chair — Faculty of Pharmacy, Pharos University, Alexandria, Egypt; Hala Abo El-hassan, Study Chair — Faculty of Pharmacy, Pharos University, Alexandria, Egypt; Ramy Elwaraky, Study Chair — Department of Clinical Pharmacy, Kidney and Urology Center, Alexandria, Egypt; Engy Emam, Study Chair — Clinical Pharmacist, Alexandria Main University Hospital, Alexandria, Egypt
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Scherberich JE, Funfstuck R, Naber KG. Urinary tract infections in patients with renal insufficiency and dialysis - epidemiology, pathogenesis, clinical symptoms, diagnosis and treatment. GMS Infect Dis. 2021 Dec 21;9:Doc07. doi: 10.3205/id000076. eCollection 2021. PMID 35106269
- [Background] Gouda Z, Mashaal G, Bello AK, El Attar A, El Kemmry T, El Reweny A, El Nahas M. Egypt Information, Prevention, and Treatment of Chronic Kidney Disease (EGIPT-CKD) programme: prevalence and risk factors for microalbuminuria among the relatives of patients with CKD in Egypt. Saudi J Kidney Dis Transpl. 2011 Sep;22(5):1055-63. PMID 21912051
- [Background] Dimitrijevic Z, Paunovic G, Tasic D, Mitic B, Basic D. Risk factors for urosepsis in chronic kidney disease patients with urinary tract infections. Sci Rep. 2021 Jul 13;11(1):14414. doi: 10.1038/s41598-021-93912-3. PMID 34257397